CLINICAL TRIAL: NCT02172794
Title: A Randomised, Double-Blind, Double-Dummy, Placebo-Controlled, Crossover Comparison of the Effect of 6-Week Treatment Periods of Tiotropium Inhalation Capsules (18 μg) and Salmeterol Inhalation Aerosol on Muscular Efficiency and Resting Energy Expenditure (REE) in Patients With Stable Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Tiotropium Inhalation Capsules and Salmeterol Inhalation Aerosol on Muscular Efficiency and Resting Energy Expenditure (REE) in Patients With Stable Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.261
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate

ARMS (2):
- tiotropium (Experimental)
  Interventions: Drug: Tiotropium; Drug: Placebo to tiotropium
- salmeterol (Active Comparator)
  Interventions: Drug: Salmeterol; Drug: Placebo to salmeterol

INTERVENTIONS:
Drug: Tiotropium
  Arms: tiotropium
Drug: Placebo to tiotropium
  Arms: tiotropium
Drug: Salmeterol
  Arms: salmeterol
Drug: Placebo to salmeterol
  Arms: salmeterol

SUMMARY:
The primary objective of this study is to evaluate the effect of tiotropium on gross muscular efficiency

ELIGIBILITY:
Inclusion Criteria:

1. All patients had to sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions.
2. Male or female patients 40 years of age or older.
3. All patients had to have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   Patients had to have moderate to severe airway obstruction with a postbronchodilator FEV1/FVC ≤ 70% and FEV1 ≤ 60% predicted (Visit 1).
4. FEV1 % predicted and/or forced vital capacity (FVC) increases >5% after inhalation with 480 μg salbutamol and 80 μg ipratropium
5. Patients had to be current or ex-smokers with a smoking history of more than 10 pack-years.
6. Patients had to be able to perform technically acceptable pulmonary function tests and had to be able to maintain records (Patient Daily Record) during the study period as required in the protocol.
7. Patients had to be able to inhale medication from the HandiHaler, and from an inhalation aerosol.
8. Patients should have had a ventilatory limitation of maximal exercise capacity:

   Increase in arterial carvon dioxide tension (PaCO2) during incremental bicycle test and/or increase in minute ventilation (VE) max > 80% (FEV1 x 37.5)
9. Patients should have had a Wmax ≥ 40 Watt during maximal incremental bicycle test.

Exclusion Criteria:

1. Increase of blood lactate > 10 mmol/L at peak exercise
2. Increase of blood lactate >2.5 mmol/L at ≥ 50% of Wmax
3. Decrease of oxygen saturation below 90% at ≥ 50% of Wmax
4. Patients with significant diseases other than COPD had to be excluded. A significant disease was defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
5. Patients with clinically relevant abnormal haemoglobulin, leukocytes, thrombocytes, glucose, sodium, potassium.
6. Patients with a recent history (i.e., six months or less) of myocardial infarction.
7. Patients with any cardiac arrhythmia requiring drug therapy or who have been hospitalised for heart failure within the past three years.
8. Patients with known active tuberculosis.
9. Patients on oxygen therapy.
10. Patients with a history of cystic fibrosis, bronchiectasis, interstitial lung disease, or pulmonary thromboembolic disease.
11. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion 4.
12. Patients with any respiratory infection in the six weeks prior to the Screening Visit (Visit 1) or during the baseline period. The enrolment of these patients was to be postponed for at least six weeks.
13. Patients who have frequent exacerbations (at least three in the preceding year) which could be expected to interfere with the patient's ability to participate in the trial should be excluded.
14. Patients with known hypersensitivity to anticholinergic drugs, beta adrenergics, lactose or any other components of the inhalation capsule delivery system.
15. Patients with a history of cancer within the last three years. Patients with treated basal cell carcinoma were allowed. Patients with successfully treated cancers greater than five years prior to entry were allowed.
16. Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction.
17. Patients with known narrow-angle glaucoma.
18. Patients who were being treated with cromolyn sodium or nedocromil sodium.
19. Patients who were being treated with antihistamines (H1 receptor antagonists).
20. Patients who were being treated with theophyllines
21. Patients who were currently on β-blocker therapy.
22. Patients using oral corticosteroid medication at unstable doses (i.e. less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
23. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception for the previous 3 months (i.e. oral contraceptives, intrauterine devices, diaphragm or subdermal implants e.g. Norplant).
24. Patients with a history of asthma or allergic rhinitis or who have a total blood eosinophil count ≥600 /mm3. A repeat eosinophil count was not conducted in these patients (Criterion modified by Protocol Amendment 2).
25. Patients with significant alcohol or drug abuse within the past two years.
26. Patients who had taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit (Visit 1).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-05; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Bruto muscular efficiency by one-point measurement of energy expenditure (EE) during bicycling at 50% Wmax | Day 42, 84, 126

SECONDARY OUTCOMES:
Resting energy expenditure (REE) | Day 42, 84, 126
Endurance capacity in minutes | Day 42, 84, 126
Nett muscular efficiency (%) | Day 42, 84, 126
Forced expiratory volume in one second (FEV1) | Up to day 140
Peak expiratory flow (PEF) variability | Up to day 140
Specific airway conductance (sGaw) | Day 42, 84, 126
Functional residual capacity (FRC) | Day 42, 84, 126
COPD Control Questionnaire (CCQ) scores on a 7 point scale | Day 42, 84, 126
Number of Participants with Adverse Events | up to day 140
Change from baseline in pulse rate | Baseline, up to day 140
Change from baseline in blood pressure | Baseline, up to day 140